CLINICAL TRIAL: NCT05818813
Title: The Long-term Safety and Effect of Renal Denervation for Resistant Hypertension
Brief Title: The Long-term Safety and Effect of Renal Denervation
Acronym: RDN flow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 14/LO/0026
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
Keywords: Hypertension; Renal denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Renal denervation — Renal denervation (ReCor Medical)

SUMMARY:
The goal of this observational study is to learn about the effects of renal denervation in patients with resistant hypertension. The main question it aims to answer is: What are the long term effects of renal denervation on blood pressure and flow within the arteries? Participants will undergo an assessment of their blood pressure, echocardiogram and invasive measurements of blood pressure and flow in the aorta and renal arteries before undergoing the renal denervation procedure. 6 months later these assessments will be repeated.

DETAILED DESCRIPTION:
Renal denervation is emerging as a succesful technique in the treatment of high blood pressure particularly for those people who's disease is resistant to drug therapy. It involves insertion of an catheter through the femoral artery and into the renal artery where it delivers a controlled radiofrequency ablation to the renal artery wall.

The purpose of this ablation is to interupt the sympathetic nervous system which is inappropriately activated in hypertension. Its beneficial effects on BP reduction has been borne out in a recently published randomised clinical trial which demonstrated a reduction in blood pressure in patients who underwent denervation compared to those managed with medication alone and it is now being used worldwide to manage hypertensive patients.

The safety of this procedure has been demonstrated in the peri-operative setting and short term particularly regarding anatomical changes and kidney function. However, its effects have not been demonstrated with invasive imaging or physiological testing in the long term. Therefore, the investigators recognise that a repeat assessment 6 months after denervation using invasive measures (to perform detailed assessments of the effects on aortic, flow and artery stiffness) would be of great benefit in stratifying this technique, which is likely to become widespread in the very near future.

The investigators therefore plan to perform denervation in 20 patients and obtain detailed information on kidney and aortic blood pressure and flow. They will then reassess these parameters after 6 months in the same patients to ensure preservation of pressure, flow and energy transfer and document the effects of denervation on vascular stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure >160mmHg despite 3 antihypertensive agents
* eGFR >45

Exclusion Criteria:

* Secondary causes of hypertension
* Prior renal artery intervention
* Renal insufficiency
* Significant stenotic valvular heart disease
* Myocardial infarction, unstable angina or stroke within the preceding 6 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with resistant hypertension and no contraindication to renal denervation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | At baseline and at 6 months
  Invasively measured aortic systolic pressure

SECONDARY OUTCOMES:
Change in diastolic pressure | At baseline and 6 months
  Invasively measured aortic diastolic pressure
Change in renal artery pressure | At baseline and 6 months
  Invasively measured
Change in renal artery flow | At baseline and 6 months
  Invasively measured
Change in renal artery resistance | At baseline and 6 months
  Invasively measured
Change in aortic reservoir pressure | At baseline and 6 months
  Invasively measured
Change in aortic wavespeed | At baseline and 6 months
  Invasively measured
Change in aortic reservoir wave intensity | At baseline and 6 months
  Invasively measured
Change in left ventricular wall thickness | At baseline and 6 months
  Assessed during echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Sayan Sen, PhD, Principal Investigator — Consultant Cardiologist
Locations (1):
- Hammersmith Hospital, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided